CLINICAL TRIAL: NCT04667442
Title: An Investigational Performance Evaluation of the Nanomix eLab® COVID-19 Rapid Antigen Panel With Samples From COVID-19 Positive and Negative Human Subjects
Brief Title: Investigational Performance Evaluation of the Nanomix eLab® COVID-19 Rapid Antigen Panel With Samples From COVID-19 Positive and Negative Human Subjects
Status: Completed | Type: Observational
Sponsor: Nanomix (Industry)
Responsible Party: Sponsor
Other Study IDs: Nanomix CVAG-202
Record Dates: First submitted 2020-12-10; First posted 2020-12-14 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Nasal sample (without cells/ RNA/DNA) will be aliquoted and stored at Sponsor for potential future analysis/ projects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- EUA RT-PCR positive
  Interventions: Diagnostic Test: Nanomix eLab® COVID-19 Rapid Antigen Panel (non-interventional)
- EUA RT-PCR negative
  Interventions: Diagnostic Test: Nanomix eLab® COVID-19 Rapid Antigen Panel (non-interventional)

INTERVENTIONS:
Diagnostic Test: Nanomix eLab® COVID-19 Rapid Antigen Panel (non-interventional) — COVID-19 Rapid Antigen Diagnostic Test

SUMMARY:
Prospective samples will be collected to evaluate the agreement between a EUA RT-PCR test as the comparator method against the Nanomix eLab® system.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Male or Female
* Willing and able to provide informed consent
* Symptomatic or asymptomatic
* The EUA RT-PCR sample must be collected within one (1) day of the sample collected for testing by the Nanomix eLab® COVID-19 Rapid Antigen Panel.

Exclusion Criteria:

* Subjects without both a valid EUA RT-PCR test result and a valid Nanomix eLab® COVID-19 Rapid Antigen results will be excluded
* Subjects not being able to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include both symptomatic and asymptomatic subjects. Although to enrich for COVID-19 positive subjects, the study will preferentially identify and enrolled subjects who have been or will be tested by EUA RT-PCR including those who are symptomatic or hospitalized with symptoms, specifically those within 7-days of symptom onset that meet the study enrollment inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Demonstrate clinical agreement between an EUA RT-PCR methodology and the Nanomix eLab® COVID-19 Rapid Antigen Panel | Up to 1 year
  An analysis of the result from subjects who have been or will be tested by EUA RT-PCR will be performed to establish the sensitivity by positive percent agreement (PPA) and the specificity by negative percent agreement (NPA) of the Nanomix eLab® COVID-19 Rapid Antigen Panel and a confirmatory EUA RT-PCR method.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Landess, Study Director — Nanomix
Locations (1):
- Nanomix, Emeryville, California, United States

IPD SHARING:
Plan to Share IPD: No